CLINICAL TRIAL: NCT00086931
Title: A Phase I/II Study of Weekly Intravenous Oxaliplatin in Combination With Oral Daily Capecitabine and Radiation Therapy in the Neoadjuvant Treatment of Rectal Cancer
Brief Title: Oxaliplatin, Capecitabine, and Radiation Therapy in Treating Patients With Locally Advanced Cancer of the Rectum
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 10803; RPCI-I-10803; SANOFI-RPCI-I-10803
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage III rectal cancer; stage II rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine — oral dose escalating, twice daily.
Drug: oxaliplatin — IV over 2 hours on days 1, 8, 15, 22, and 29.
Procedure: conventional surgery — curative-intent surgery 6-8 weeks after the completion of chemoradiotherapy
Procedure: neoadjuvant therapy — chemotherapy and radiation prior to surgery
Radiation: radiation therapy — once daily 5 days a week for 5.5 weeks

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin and capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Oxaliplatin and capecitabine may make tumor cells more sensitive to radiation therapy and may kill more tumor cells. Giving chemotherapy with radiation therapy before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase I/II trial is studying the side effects and best dose of oxaliplatin and capecitabine when given together with radiation therapy and to see how well they work in treating patients who are undergoing surgery for locally advanced cancer of the rectum. NOTE: *The phase I portion of this trial closed 06/2005. The best dose of oxaliplatin and capecitabine has been determined.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of neoadjuvant oxaliplatin and capecitabine when combined with radiotherapy in patients with locally advanced adenocarcinoma of the rectum. (Phase I closed to accrual as of 06/2005.)
* Determine the rate of complete pathological response in patients treated with this regimen.

Secondary

* Determine the overall survival of patients treated with this regimen.
* Determine the rate of local and overall failure in patients treated with this regimen.
* Determine the utility of TS, TP, DPD, ERCC-1, and apoptosis to predict response in patients treated with this regimen.
* Determine the rate of pathologic down-staging in patients treated with this regimen.
* Determine the safety and toxicity of this regimen in these patients.
* Determine the rate of sphincter-saving rectal surgery in patients treated with this regimen who had been deemed candidates for abdominoperineal resection at diagnosis.

OUTLINE: This is a multicenter, phase I (phase I closed to accrual as of 06/2005), dose-escalation study of oxaliplatin and capecitabine followed by a phase II study.

* Phase I (closed to accrual as of 06/2005): Patients undergo radiotherapy once daily 5 days a week for 5.5 weeks and receive oral capecitabine twice daily on days radiotherapy is administered. Beginning on day 1 of radiotherapy, patients also receive oxaliplatin IV over 2 hours on days 1, 8, 15, 22, and 29.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients undergo radiotherapy and receive capecitabine and oxaliplatin as in phase I at the MTD.

All patients undergo curative-intent surgery 6-8 weeks after the completion of chemoradiotherapy.

Patients are followed every 3 months for 3 years and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 31-40 patients (6-15 for phase I [phase I closed to accrual as of 06/2005] and 25 for phase II) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * Tumor involving the distal 12 cm of the rectum (above the anal verge)
  * Clinically staged by endoscopic ultrasound with one of the following criteria:

    * T3-T4 disease
    * Evidence of lymph node involvement, defined by the presence of ≥ 1 enlarged peri-rectal lymph node (≥ 1 cm in size)
* No known distant metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* ECOG 0-1 OR
* Karnofsky 70-100%

Life expectancy

* More than 1 year

Hematopoietic

* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Able to receive oral medication
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No prior or concurrent significant neuropathy
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study drugs
* No ongoing or active infection
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent granulocyte-stimulating factors

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic radiotherapy

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2003-09; Primary Completion 2007-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Complete pathological response rate at time of surgery | Time of surgery

SECONDARY OUTCOMES:
Disease-free survival, safety, and overall survival at 5 years | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Fakih MG, Bullarddunn K, Yang GY, Pendyala L, Toth K, Andrews C, Rustum YM, Ross ME, Levea C, Puthillath A, Park YM, Rajput A. Phase II study of weekly intravenous oxaliplatin combined with oral daily capecitabine and radiotherapy with biologic correlates in neoadjuvant treatment of rectal adenocarcinoma. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):650-7. doi: 10.1016/j.ijrobp.2008.01.020. Epub 2008 Jun 17. PMID 18565686
- [Result] Fakih MG, Rajput A, Yang GY, et al.: A phase I and biological correlates study of capecitabine (CAP) + oxaliplatin (OX) + radiation therapy (RT) in locally advanced rectal cancer (LARC). [Abstract] J Clin Oncol 23 (Suppl 16): A-3633, 279s, 2005.